CLINICAL TRIAL: NCT02807519
Title: Salivary Cytokines in Paediatric Oncology Patients and Healthy Persons - A Pilot Study to Investigation of Biomarkers for Oral Health
Brief Title: Salivary Cytokines as Biomarker for Oral Health
Acronym: Cytosal
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Schulzahnklinik Basel (Unknown); Volkszahnklinik Basel (Unknown)
Responsible Party: Sponsor
Other Study IDs: UKBB-2016/011
Record Dates: First submitted 2016-06-13; First posted 2016-06-21 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Neoplasms
Keywords: Oral health; Saliva; Biomarker; Cytokines; Cancer; children
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva sample collection. Cytokines analysis in the saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Oncological patients: Children with confirmed haematological/oncological diagnosis who are admitted to the paediatric oncology ward at the Universitätsspital Beider Basel (UKBB), who will require radio- and/or chemotherapy . Collection of salivary cytokines will be performed in this group.
  Interventions: Genetic: collection of salivary cytokines
- Control group: Healthy children which are seen routinely at the Schulzahnklinik/Volkzahnklinik Basel. Collection of salivary cytokines will be performed in this group.
  Interventions: Genetic: collection of salivary cytokines

INTERVENTIONS:
Genetic: collection of salivary cytokines — Collection of the saliva will be done following this procedure: The collection will be done prior to any other dental manipulation. The test person is sitting with its head tilted slightly forward. Initially, any saliva present in the mouth must be swallowed or spit out completely. Then, a paraffin gum is given to the test person. This paraffin gum must be chewed for minimally 2 and maximally up to 5 minutes. During the time period that the test person is chewing the paraffin gum, the saliva must be spitted into a cup repeatedly, or the saliva can also be let run passively into the cup. The amount of saliva is then weighted (1g equivalent to 1 ml) and a saliva flow rate (ml/min) is calculated and noted.

SUMMARY:
Oral complications during and after cancer treatment are common. A key role in maintaining oral health plays saliva. In the last decade numerous studies have investigated immunological biomarkers such as cytokines in saliva samples. In children, the few studies have investigated salivary cytokines (sCK) suggesting that these are associated with oral health (sCK). One study investigating sCK in adult oncology patients showed an association between Interleukin-6 (IL-6) and severity of oral chronic graft-versus-host disease (GVHD) in survivors of hematopoietic stem cell transplantation. Therefore determination of sCK concentrations may also be helpful for assessment of GVHD activity and other inflammatory processes in cancer patients. In pediatric oncology patients, to the investigators' knowledge, no study has so far investigated sCK concentrations as markers for oral or systemic health.

DETAILED DESCRIPTION:
Oral complications are common during and after cancer treatment. Oral mucositis typically occurs during or immediately after chemotherapy and may lead to pain, oral and systemic infection, and nutritional compromise. Late effects of oral mucositis as a result of cancer treatment include an increased risk for dental caries, xerostomia and osteonecrosis. It has been recognised, that regular assessment of oral health, prevention and early treatment of oral mucositis decreases early and late complication rates.

Saliva plays a key role in maintaining oral health and reduced salivary flow contributes to acute disorders and long-term sequelae in oral health. Saliva is a complex fluid secreted by the salivary glands and the gingiva. In the last decade numerous studies have investigated immunological biomarkers such as cytokines in saliva samples. These studies included individuals with various oral and systemic diseases including oral cancer, oral caries, autoimmune and endocrine diseases, metabolic syndrome, chronic kidney disease and psychiatric illnesses.

In children, the few studies that have investigated salivary cytokines (sCK) suggest that these are associated with oral health (sCK). For example, one study in 114 healthy adolescent girls aged 11-17 years showed that sCK concentrations were generally not associated with levels in the serum . In addition this study also suggested that the sCK concentrations are age dependent.

However, a number of other studies suggest that sCK may also reflect systemic diseases such as shown in a study including 20 children aged 9-17 with allergies (including asthma, allergic rhinitis and eosinophilic esophagitis) showing that Th-2 cytokines were detectable in sCK.

One study investigating sCK in adult oncology patients showed an association between IL-6 and severity of oral chronic GVHD in survivors of a hematopoietic stem cell transplantation. Therefore determination of sCK concentrations may also be helpful for assessment of GVHD activity and other inflammatory processes in cancer patients. In paediatric oncology patients, to the investigators' knowledge, no study has so far investigated sCK concentrations as markers for oral or systemic health.

ELIGIBILITY:
Inclusion Criteria:

* Children with confirmed haematological/oncological disease and necessity for radio-or chemotherapy
* Age > 4 and < 18 years.

Exclusion Criteria:

* patients, who already were treated with radio- or chemotherapy
* patients with current or previous (last 7 days) symptoms of a respiratory infection, rhinitis, bronchitis and tonsillitis
* children with an autoimmune disease
* Use of systemic antibiotics within the last 2 weeks.
* Use of antimicrobial mouth rinsing solution within the last 12 hours,
* any vaccination within the last 48 hours
* known allergy to paraffin.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: * Children with a new haematological/oncological diagnosis
  * admitted to the paediatric oncology ward at the UKBB
  * who will require radio- and/or chemotherapy.
  Healthy children who present at the Schulzahnklinik respectively Volkszahnklinik for a dental prophylaxis
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
mucositis (clinical oral finding) | 18 months
  clinical oral finding as mucositis in children with a hematological/oncological disease and healthy control children
salivary cytokine (sCK) levels | 18 months
  salivary cytokine (sCK) levels in children with a hematological/oncological disease and healthy control children
aphthous ulcer (clinical oral finding) | 18 months
  clinical oral finding as aphthous ulcer in children with a hematological/oncological disease and healthy control children

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Diesch, Dr., Principal Investigator — University Children's Hospital of Basel; Cornelia Filippi, Dr., Principal Investigator — University Centre of Dental Medicine Basel
Locations (3):
- Switzerland (3):
  - Schulzahlklinik Basel, Basel, Canton of Basel-City
  - Volkszahnklinik, Basel, Canton of Basel-City
  - Kinderspital Aarau, Aarau

IPD SHARING:
Plan to Share IPD: Undecided